CLINICAL TRIAL: NCT03758443
Title: A Phase 2b/3 Multi-Center, Randomized, Double-Blind, Multi-Dose, Placebo-Controlled, Parallel-Group Set of Studies to Evaluate the Efficacy and Safety of Induction and Maintenance Therapy With TD-1473 in Subjects With Moderately-to-Severely Active Ulcerative Colitis
Brief Title: Efficacy & Safety of TD-1473 in Ulcerative Colitis
Acronym: RHEA
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Stopped early due to company decision. Company decision based on interim analysis results in TD-1473-0157.
Sponsor: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0157; 2018-002136-24 (EudraCT Number)
Record Dates: First submitted 2018-11-19; First posted 2018-11-29 (Actual); Results first posted 2022-11-15 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2021-11

CONDITIONS: Ulcerative Colitis (UC)
Keywords: TD-1473; Janus kinase inhibitor; JAK inhibitor; Inflammatory Bowel Disease; IBD; Ulcerative colitis; UC; Gut selective
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: Integrated and Adaptive Design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Active Treatment TD-1473 Dose A (Experimental): Participants will be randomized to receive an oral daily dose of TD-1473. Responders will be re-randomized into the Phase 3 Maintenance portion of the study. Non-responders may participate in an extended induction.
  Interventions: Drug: TD-1473 Dose A
- Active Treatment TD-1473 Dose B (Experimental): Participants will be randomized to receive an oral daily dose of TD-1473. Responders will be re-randomized into the Phase 3 Maintenance portion of the study. Non-responders may participate in an extended induction.
  Interventions: Drug: TD-1473 Dose B
- Active Treatment TD-1473 Dose C (Experimental): Participants will be randomized to receive an oral daily dose of TD-1473. Responders will be re-randomized into the Phase 3 Maintenance portion of the study. Non-responders may participate in an extended induction.
  Interventions: Drug: TD-1473 Dose C
- Placebo (Placebo Comparator): Participants will be randomized to receive an oral daily dose of placebo. Participants who received Placebo (and were non-responders) may move to an extended induction. Subjects who are on placebo will be assigned to active TD-1473 for the extended induction (they will be blinded to dose).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TD-1473 Dose A — See Arm description
  Arms: Active Treatment TD-1473 Dose A
Drug: TD-1473 Dose B — See Arm description
  Arms: Active Treatment TD-1473 Dose B
Drug: TD-1473 Dose C — See Arm description
  Arms: Active Treatment TD-1473 Dose C
Drug: Placebo — See Arm description
  Arms: Placebo

SUMMARY:
A Phase 2b/3 set of studies to evaluate the efficacy and safety of induction and maintenance therapy with TD-1473 in subjects with moderately-to-severely active ulcerative colitis with up to 60 weeks of treatment.

DETAILED DESCRIPTION:
This protocol consists of 3 separate studies: an 8-week Phase 2b dose-finding induction study, an 8-week dose-confirming Phase 3 induction study, and a 44-week Phase 3 maintenance study. Subjects who respond to induction will enter the maintenance study; those who do not will receive TD-1473 during extended induction. The safety and efficacy data of the Phase 2b study will be analyzed to select the induction and maintenance dose regimens for the confirmatory Phase 3 studies. Participants who have disease relapse or complete the maintenance study may be eligible to enter a separate long-term safety study. Efficacy, pharmacokinetic, biomarkers, and safety will be evaluated in all 3 studies.

240 subjects are planned for the Phase 2b and the planned Primary Completion Date for this portion of the study is JULY 2021. 640 subjects are planned for the Phase 3 portion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 18 years of age at screening
* Has a history of UC for at least 3 months prior to screening
* Has moderately-to-severely active UC, as defined by a Mayo endoscopic subscore of ≥2 points and an adapted Mayo score between 4 - 9 points inclusive
* Is corticosteroid-dependent or has demonstrated inadequate response, or intolerance to conventional therapy (aminosalicylates, corticosteroids, immunomodulators) or biologics
* Willing to use highly-effective methods of contraception during the study and for 7 days after the last dose
* Additional inclusion criteria apply

Exclusion Criteria:

* Has symptoms suggestive of fulminant colitis, megacolon or intestinal perforation
* Likely to require surgery for UC or other major surgeries
* Has previously received / is currently receiving prohibited medications within specified timeframe
* Is refractory to 3 biologics with ≥2 mechanisms of action
* Has a current bacterial, parasitic, fungal, or viral infection
* Has clinically significant abnormalities in laboratory evaluations
* Has had any prior exposure to an approved Janus kinase (JAK) inhibitor or potential exposure to an investigational JAK inhibitor that was stopped due to intolerance or lack of efficacy
* Additional exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 239 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2021-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (165):
- United States (37):
  - Theravance Biopharma Investigational Site, Chula Vista, California
  - Theravance Biopharma Investigational Site, La Jolla, California
  - Theravance Biopharma Investigational Site, Lancaster, California
  - Theravance Biopharma Investigational Site, Orange, California
  - Theravance Biopharma Investigational Site, Colorado Springs, Colorado
  - Theravance Biopharma Investigational Site, Aventura, Florida
  - Theravance Biopharma Investigational Site, Clearwater, Florida
  - Theravance Biopharma Investigational Site, Largo, Florida
  - Theravance Biopharma Investigational Site, Miami, Florida
  - Theravance Biopharma Investigational Site, New Port Richey, Florida
  - Theravance Biopharma Investigational Site, New Smyrna Beach, Florida
  - Theravance Biopharma Investigational Site, Orlando, Florida
  - Theravance Biopharma Investigational Site, Pembroke Pines, Florida
  - Theravance Biopharma Investigational Site, Atlanta, Georgia
  - Theravance Biopharma Investigational Site, Suwanee, Georgia
  - Theravance Biopharma Investigational Site, Idaho Falls, Idaho
  - Theravance Biopharma Investigational Site, Kansas City, Kansas
  - Theravance Biopharma Investigational Site, Louisville, Kentucky
  - Theravance Biopharma Investigational Site, Monroe, Louisiana
  - Theravance Biopharma Investigational Site, Baltimore, Maryland
  - Theravance Biopharma Investigational Site, Troy, Michigan
  - Theravance Biopharma Investigational Site, Wyoming, Michigan
  - Theravance Biopharma Investigational Site, Rochester, Minnesota
  - Theravance Biopharma Investigational Site, Kansas City, Missouri
  - Theravance Biopharma Investigational Site, Las Vegas, Nevada
  - Theravance Biopharma Investigational Site, New York, New York
  - Theravance Biopharma Investigational Site, Charlotte, North Carolina
  - Theravance Biopharma Investigational Site, Gastonia, North Carolina
  - Theravance Biopharma Investigational Site, Greenville, North Carolina
  - Theravance Biopharma Investigational Site, Pittsburgh, Pennsylvania
  - Theravance Biopharma Investigational Site, Smithfield, Pennsylvania
  - Theravance Biopharma Investigational Site, Greenville, South Carolina
  - Theravance Biopharma Investigational Site, Rock Hill, South Carolina
  - Theravance Biopharma Investigational Site, Nashville, Tennessee
  - Theravance Biopharma Investigational Site, Garland, Texas
  - Theravance Biopharma Investigational Site, Houston, Texas
  - Theravance Biopharma Investigational Site, San Antonio, Texas
- Australia (4):
  - Theravance Biopharma Investigational Site, South Brisbane, Queensland
  - Theravance Biopharma Investigational Site, Woolloongabba, Queensland
  - Theravance Biopharma Investigational Site, Malvern, Victoria
  - Theravance Biopharma Investigational Site, Murdoch, Western Australia
- Bulgaria (9):
  - Theravance Biopharma Investigational Site, Sofia, Sofia
  - Theravance Biopharma Investigational Site (2), Pleven
  - Theravance Biopharma Investigational Site, Pleven
  - Theravance Biopharma Investigational Site, Plovdiv
  - Theravance Biopharma Investigational Site, Rousse
  - Theravance Biopharma Investigational Site, Sliven
  - Theravance Biopharma Investigational Site, Sofia
  - Theravance Biopharma Investigational Site, Stara Zagora
  - Theravance Biopharma Investigational Site, Veliko Tarnovo
- Theravance Biopharma Investigational Site, Kingston, Ontario, Canada
- France (9):
  - Theravance Biopharma Investigational Site, Pierre-Bénite, Auvergne-Rhône-Alpes
  - Theravance Biopharma Investigational Site, Saint-Etienne, Auvergne-Rhône-Alpes
  - Theravance Biopharma Investigational Site, Reims, Champagne-ardenne
  - Theravance Biopharma Investigational Site, Lille, Hauts-de-France
  - Theravance Biopharma Investigational Site, Montpellier, Languedoc-roussillon
  - Theravance Biopharma Investigational Site, Vandœuvre-lès-Nancy, Limousin
  - Theravance Biopharma Investigational Site, Toulouse, Midi-pyrenees
  - Theravance Biopharma Investigational Site, Nantes, Pays de la Loire Region
  - Theravance Biopharma Investigational Site, Amiens, Picardie
- Georgia (2):
  - Theravance Biopharma Investigational Site, Batumi
  - Theravance Biopharma Investigational Site, Tbilisi
- Germany (5):
  - Theravance Biopharma Investigational Site, Heidelberg, Baden-Wurttemberg
  - Theravance Biopharma Investigational Site, Ulm, Baden-Wurttemberg
  - Theravance Biopharma Investigational Site, Kiel, Schleswig-Holstein
  - Theravance Biopharma Investigational Site, Jena, Thuringia
  - Theravance Biopharma Investigational Site, Berlin
- Greece (4):
  - Theravance Biopharma Investigational Site, Athens, Attica
  - Theravance Biopharma Investigational Site #2, Athens, Attica
  - Theravance Biopharma Investigational Site, Heraklion, Crete
  - Theravance Biopharma Investigational Site, Patra, Peloponnese
- Hungary (4):
  - Theravance Biopharma Investigational Site, Székesfehérvár, Fejér
  - Theravance Biopharma Investigational Site, Debrecen, Hajdú-Bihar
  - Theravance Biopharma Investigational Site, Szekszárd, Tolna County
  - Theravance Biopharma Investigational Site, Budapest
- Israel (7):
  - Theravance Biopharma Investigational Site, Ẕerifin, Rehoboth
  - Theravance Biopharma Investigational Site, Haifa
  - Theravance Biopharma Investigational Site, Holon
  - Theravance Biopharma Investigational Site, Jerusalem
  - Theravance Biopharma Investigational Site, Nahariya
  - Theravance Biopharma Investigational Site, Petah Tikva
  - Theravance Biopharma Investigational Site, Rehovot
- Italy (3):
  - Theravance Biopharma Investigational Site, Rozzano, Milano
  - Theravance Biopharma Investigational Site, Catanzaro
  - Theravance Biopharma Investigational Site, Pavia
- Japan (21):
  - Theravance Biopharma Investigational Site, Nagoya, Aichi-ken
  - Theravance Biopharma Investigational Site, Abiko, Chiba
  - Theravance Biopharma Investigational Site, Sakura, Chiba
  - Theravance Biopharma Investigational Site, Kurume, Fukuoka
  - Theravance Biopharma Investigational Site, Ōgaki, Gifu
  - Theravance Biopharma Investigational Site, Isesaki, Gunma
  - Theravance Biopharma Investigational Site, Fukuyama-Shi, Hiroshima
  - Theravance Biopharma Investigational Site, Hatsukaichi, Hiroshima
  - Theravance Biopharma Investigational Site, Kawasaki, Kanagawa
  - Theravance Biopharma Investigational Site, Sendai, Miyagi
  - Theravance Biopharma Investigational Site, Suwa, Nagano
  - Theravance Biopharma Investigational Site, Ōita, Oita Prefecture
  - Theravance Biopharma Investigational Site, Fujiidera, Osaka
  - Theravance Biopharma Investigational Site, Izumiōtsu, Osaka
  - Theravance Biopharma Investigational Site, Ageo, Saitama
  - Theravance Biopharma Investigational Site, Tokorozawa, Saitama
  - Theravance Biopharma Investigational Site, Kurobe-shi, Toyama
  - Theravance Biopharma Investigational Site, Chiba
  - Theravance Biopharma Investigational Site, Fukuoka
  - Theravance Biopharma Investigational Site, Kumamoto
  - Theravance Biopharma Investigational Site, Tokyo
- Poland (15):
  - Theravance Biopharma Investigational Site, Poznan, Greater Poland Voivodeship
  - Theravance Biopharma Investigational Site, Torun, Kuyavian-Pomeranian Voivodeship
  - Theravance Biopharma Investigational Site, Włocławek, Kuyavian-Pomeranian Voivodeship
  - Theravance Biopharma Investigational Site, Krakow, Lesser Poland Voivodeship
  - Theravance Biopharma Investigational Site, Lodz, Lodzki
  - Theravance Biopharma Investigational Site, Wroclaw, Lower Silesian Voivodeship
  - Theravance Biopharma Investigational Site, Piaseczno, Masovian Voivodeship
  - Theravance Biopharma Investigational Site, Warsaw, Masovian Voivodeship
  - Theravance Biopharma Investigational Site, Sopot, Pomeranian Voivodeship
  - Theravance Biopharma Investigational Site, Tychy, Silesian Voivodeship
  - Theravance Biopharma Investigational Site, Szczecin, West Pomeranian Voivodeship
  - Theravance Biopharma Investigational Site, Szczecin
  - Theravance Biopharma Investigational Site, Ksawerów, Łódź Voivodeship
  - Theravance Biopharma Investigational Site, Lodz, Łódź Voivodeship
  - Theravance Biopharma Investigational Site, Staszów, Świętokrzyskie Voivodeship
- Portugal (8):
  - Theravance Biopharma Investigational Site, Coimbra
  - Theravance Biopharma Investigational Site, Guimarães
  - Theravance Biopharma Investigational Site, Leiria
  - Theravance Biopharma Investigational Site, Lisbon
  - Theravance Biopharma Investigational Site, Santa Maria da Feira
  - Theravance Biopharma Investigational Site, Senhora da Hora
  - Theravance Biopharma Investigational Site, Viana do Castelo
  - Theravance Biopharma Investigational Site, Vila Nova de Gaia
- Romania (2):
  - Theravance Biopharma Investigational Site, Timișoara, Timiș County
  - Theravance Biopharma Investigational Site, Bucharest
- Serbia (5):
  - Theravance Biopharma Investigational Site, Belgrade
  - Theravance Biopharma Investigational Site, Kragujevac
  - Theravance Biopharma Investigational Site, Niš
  - Theravance Biopharma Investigational Site, Subotica
  - Theravance Biopharma Investigational Site, Zrenjanin
- Slovakia (3):
  - Theravance Biopharma Investigational Site, Prešov, Prešovsky
  - Theravance Biopharma Investigational Site, Nitra
  - Theravance Biopharma Investigational Site, Šahy
- Theravance Biopharma Investigational Site, Johannesburg, Gauteng, South Africa
- South Korea (4):
  - Theravance Biopharma Investigational Site, Wŏnju, Gangwon-do
  - Theravance Biopharma Investigational Site, Suwon, Gyeonggi-do
  - Theravance Biopharma Investigational Site, Daegu
  - Theravance Biopharma Investigational Site, Seoul
- Spain (4):
  - Theravance Biopharma Investigational Site, Barcelona
  - Theravance Biopharma Investigational Site, Madrid
  - Theravance Biopharma Investigational Site, Seville
  - Theravance Biopharma Investigational Site, Valencia
- Taiwan (4):
  - Theravance Biopharma Investigational Site, Kaohsiung City
  - Theravance Biopharma Investigational Site, Taichung
  - Theravance Biopharma Investigational Site, Tainan
  - Theravance Biopharma Investigational Site, Taipei
- Ukraine (13):
  - Theravance Biopharma Investigational Site, Kiev, KIEV CITY
  - Theravance Biopharma Investigational Site, Kyiv, Kyiv City
  - Theravance Biopharma Investigational Site, Kremenchuk, Poltava Oblast
  - Theravance Biopharma Investigational Site, Uzhhorod, Transcarpathian
  - Theravance Biopharma Investigational Site, Vinnytsia, Vinnytsya
  - Theravance Biopharma Investigational Site, Chernivtsi
  - Theravance Biopharma Investigational Site, Kharkiv
  - Theravance Biopharma Investigational Site #2, Lviv
  - Theravance Biopharma Investigational Site, Lviv
  - Theravance Biopharma Investigational Site, Ternopil
  - Theravance Biopharma Investigational Site, Uzhhorod
  - Theravance Biopharma Investigational Site, Vinnytsia
  - Theravance Biopharma Investigational Site, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: No
Theravance Biopharma, Inc. will not be sharing individual de-identified participant data or other relevant study documents.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 239 participants were enrolled at sites in Europe, Asia/Pacific, the United States, Israel, Australia, and South Africa between 11 March 2019 and 20 October 2021.
Groups:
- Placebo: Participants were randomized to receive once-daily administrations of placebo for 8 weeks during the Induction Period.
  Participants who achieved clinical response by adapted Mayo Score at Week 8 continued to receive blinded placebo in the Maintenance Period. Participants who did not achieve clinical response at Week 8 received 80 mg TD-1473 for 8 weeks in the Extended Induction Period.
  Participants who achieved clinical response to a total of 8 weeks of TD-1473 induction therapy, either at Week 8 or Week 16, were re-randomized to received placebo; 20 mg, 80 mg, or 200 mg TD-1473 for 44 weeks in the Maintenance Period. Participants who did not achieve clinical response to a total of 8 weeks of TD-1473 induction therapy underwent study exit procedures.
- TD-1473 20 mg: Participants were randomized to receive once-daily administrations of 20 mg TD-1473 for 8 weeks during the Induction Period.
  Participants who achieved clinical response by adapted Mayo Score at Week 8 continued to receive 20 mg TD-1473 in the Maintenance Period. Participants who did not achieve clinical response at Week 8 continued to receive 20 mg TD-1473 for 8 weeks in the Extended Induction Period.
  Participants who achieved clinical response to a total of 16 weeks of TD-1473 induction therapy continued to receive 20 mg TD-1473 for 44 weeks in the Maintenance Period. Participants who did not achieve clinical response to a total of 16 weeks of TD-1473 induction therapy underwent study exit procedures.
- TD-1473 80 mg: Participants were randomized to receive once-daily administrations of 80 mg TD-1473 for 8 weeks during the Induction Period.
  Participants who achieved clinical response by adapted Mayo Score at Week 8 continued to receive 80 mg TD-1473 in the Maintenance Period. Participants who did not achieve clinical response at Week 8 continued to receive 80 mg TD-1473 for 8 weeks in the Extended Induction Period.
  Participants who achieved clinical response to a total of 16 weeks of TD-1473 induction therapy continued to receive 80 mg TD-1473 for 44 weeks in the Maintenance Period. Participants who did not achieve clinical response to a total of 16 weeks of TD-1473 induction therapy underwent study exit procedures.
- TD-1473 200 mg: Participants were randomized to receive once-daily administrations of 200 mg TD-1473 for 8 weeks during the Induction Period.
  Participants who achieved clinical response by adapted Mayo Score at Week 8 continued to receive 200 mg TD-1473 in the Maintenance Period. Participants who did not achieve clinical response at Week 8 continued to receive 200 mg TD-1473 for 8 weeks in the Extended Induction Period.
  Participants who achieved clinical response to a total of 16 weeks of TD-1473 induction therapy continued to receive 200 mg TD-1473 for 44 weeks in the Maintenance Period. Participants who did not achieve clinical response to a total of 16 weeks of TD-1473 induction therapy underwent study exit procedures.
Period: Induction Period
Arm/Group | Placebo | TD-1473 20 mg | TD-1473 80 mg | TD-1473 200 mg
Started | 61 | 61 | 59 | 58
Completed | 55 | 54 | 52 | 50
Not Completed | 6 | 7 | 7 | 8
Not completed — Adverse Event | 2 | 4 | 2 | 3
Not completed — Physician Decision | 1 | 1 | 3 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 2 | 2 | 4
Period: Extended Induction Period
Arm/Group | Placebo | TD-1473 20 mg | TD-1473 80 mg | TD-1473 200 mg
Started | 42 (Included only participants who did not achieve clinical response at Week 8.) | 32 (Included only participants who did not achieve clinical response at Week 8.) | 32 (Included only participants who did not achieve clinical response at Week 8.) | 29 (Included only participants who did not achieve clinical response at Week 8.)
Completed | 29 | 29 | 23 | 22
Not Completed | 13 | 3 | 9 | 7
Not completed — Adverse Event | 1 | 1 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Physician Decision | 2 | 1 | 2 | 2
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 8 | 1 | 7 | 3
Not completed — Miscellaneous | 1 | 0 | 0 | 0
Period: Maintenance Period
Arm/Group | Placebo | TD-1473 20 mg | TD-1473 80 mg | TD-1473 200 mg
Started | 29 (Included only participants who achieved clinical response at Week 8 or Week 16.) | 31 (Included only participants who achieved clinical response at Week 8 or Week 16.) | 25 (Included only participants who achieved clinical response at Week 8 or Week 16.) | 22 (Included only participants who achieved clinical response at Week 8 or Week 16.)
Completed | 13 | 11 | 12 | 9
Not Completed | 16 | 20 | 13 | 13
Not completed — Adverse Event | 1 | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Persistent Loss of Response During Maintenance | 3 | 1 | 2 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Study Terminated by Sponsor | 11 | 16 | 9 | 11
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 1
Not completed — Miscellaneous | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Intent-to-treat population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | TD-1473 20 mg | TD-1473 80 mg | TD-1473 200 mg | Total
Number analyzed (Participants) | 61 | 61 | 59 | 58 | 239
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.92 (15.390) | 38.87 (14.576) | 42.02 (15.317) | 44.38 (14.122) | 41.51 (14.905)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 17 | 20 | 29 | 93
  Male | 34 | 44 | 39 | 29 | 146
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 1 | 1 | 7
  Not Hispanic or Latino | 54 | 59 | 56 | 55 | 224
  Unknown or Not Reported | 4 | 0 | 2 | 2 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 48 | 50 | 51 | 51 | 200
  Black or African American | 1 | 0 | 0 | 0 | 1
  Asian | 9 | 11 | 6 | 6 | 32
  Other | 3 | 0 | 2 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Mayo Score (tMS) at Week 8
Description: Total Mayo Score (tMS) was calculated as the sum of four components: rectal bleeding (0-3), stool frequency (0-3), physician's global assessment (0-3) and Mayo endoscopic subscore (0-3). tMS was reported as a 0-12 point score with 12 reflecting the highest severity.
Time Frame: Baseline to Week 8
Population: Modified Intent-to-Treat (mITT) Analysis Set (Induction Period): Comprised all randomized participants who received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Induction Period: Placebo: Participants were randomized to receive once-daily administrations of placebo for 8 weeks during the Induction Period.
- Induction Period: TD-1473 20 mg: Participants were randomized to receive once-daily administrations of 20 mg TD-1473 for 8 weeks during the Induction Period.
- Induction Period: TD-1473 80 mg: Participants were randomized to receive once-daily administrations of 80 mg TD-1473 for 8 weeks during the Induction Period.
- Induction Period: TD-1473 200 mg: Participants were randomized to receive once-daily administrations of 200 mg TD-1473 for 8 weeks during the Induction Period.
Arm/Group | Induction Period: Placebo | Induction Period: TD-1473 20 mg | Induction Period: TD-1473 80 mg | Induction Period: TD-1473 200 mg
Number analyzed (Participants) | 56 | 54 | 53 | 55
score on a scale | -1.75 (0.341) | -2.02 (0.350) | -2.12 (0.351) | -2.40 (0.346)
Statistical Analysis 1: Comparison: Induction Period: Placebo vs Induction Period: TD-1473 20 mg; Least square estimates, 95% CI, and p-values were obtained by fitting an ANCOVA model with terms for treatment, steroid use at baseline (yes, no) and prior biologic failure (yes, no), and baseline total Mayo score as covariate; Test type: Superiority; p = 0.5809, ANCOVA; Least Square Mean Difference = -0.27, 95% CI 2-sided [-1.22 to 0.69]
Statistical Analysis 2: Comparison: Induction Period: Placebo vs Induction Period: TD-1473 80 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.4501, ANCOVA; Least Square Mean Difference = -0.37, 95% CI 2-sided [-1.33 to 0.59]
Statistical Analysis 3: Comparison: Induction Period: Placebo vs Induction Period: TD-1473 200 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.1809, ANCOVA; Least Square Mean Difference = -0.65, 95% CI 2-sided [-1.60 to 0.30]

2. Primary Outcome: Phase 3 Maintenance: Number of Participants Who Demonstrated Clinical Remission by Adapted Mayo Score Components at Maintenance Week (mWeek) 44
Description: Clinical remission by Adapted Mayo score was defined based on Adapted Mayo score components within specific ranges: stool frequency score of 0 or 1, a rectal bleeding subscore of 0 and a Mayo endoscopy subscore of 0 or 1.
  The Adapted Mayo score was the sum of three components: rectal bleeding, stool frequency, and Mayo endoscopic subscore, each measured on a scale of 0-3 with higher scores reflecting higher severity.
  Participants with missing Week 44 values were imputed as non-responders.
Time Frame: mWeek 44
Population: mITT Analysis Set (Maintenance Period): All participants randomized into the Phase 3 Maintenance Study who were also treated. Only participants randomized at least 44 weeks prior to database lock were included.
Measure: Count of Participants; unit: Participants
Groups:
- Maintenance Period: Placebo: Participants who were randomized to receive once-daily administrations of placebo for 8 weeks during the Induction Period and achieved clinical response by adapted Mayo Score at Week 8 of the Induction Period continued to receive blinded placebo for 44 weeks in the Maintenance Period.
- Maintenance Period: TD-1473 20 mg: Participants who achieved clinical response to a total of 8 weeks of TD-1473 induction therapy, either at Week 8 or Week 16, and continued to receive 20 mg TD-1473 for 44 weeks in the Maintenance Period.
- Maintenance Period: TD-1473 80 mg: Participants who achieved clinical response to a total of 8 weeks of TD-1473 induction therapy, either at Week 8 or Week 16, and continued to receive 80 mg TD-1473 for 44 weeks in the Maintenance Period.
- Maintenance Period: TD-1473 200 mg: Participants who achieved clinical response to a total of 8 weeks of TD-1473 induction therapy, either at Week 8 or Week 16, and continued to receive 200 mg TD-1473 for 44 weeks in the Maintenance Period.
Arm/Group | Maintenance Period: Placebo | Maintenance Period: TD-1473 20 mg | Maintenance Period: TD-1473 80 mg | Maintenance Period: TD-1473 200 mg
Number analyzed (Participants) | 9 | 13 | 11 | 8
Participants | 4 | 3 | 5 | 3
Statistical Analysis 1: Comparison: Maintenance Period: Placebo vs Maintenance Period: TD-1473 20 mg; Test type: Superiority; p = 0.3762, Fisher Exact
Statistical Analysis 2: Comparison: Maintenance Period: Placebo vs Maintenance Period: TD-1473 80 mg; Test type: Superiority; p = 1.0000, Fisher Exact
Statistical Analysis 3: Comparison: Maintenance Period: Placebo vs Maintenance Period: TD-1473 200 mg; Test type: Superiority; p = 1.0000, Fisher Exact

3. Secondary Outcome: Number of Participants Who Demonstrated Clinical Remission by Adapted Mayo Score Components at Week 8
Description: Clinical remission by Adapted Mayo score was defined based on Adapted Mayo score components within specific ranges: stool frequency score of 0 or 1, a rectal bleeding subscore of 0 and a Mayo endoscopy subscore of 0 or 1.
  The Adapted Mayo score was the sum of three components: rectal bleeding, stool frequency, and Mayo endoscopic subscore, each measured on a scale of 0-3 with higher scores reflecting higher severity.
Time Frame: Week 8
Population: mITT Analysis Set (Induction Period): Comprised all randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Period: Placebo | Induction Period: TD-1473 20 mg | Induction Period: TD-1473 80 mg | Induction Period: TD-1473 200 mg
Number analyzed (Participants) | 61 | 61 | 59 | 58
Participants | 6 | 6 | 4 | 4
Statistical Analysis 1: Comparison: Induction Period: Placebo vs Induction Period: TD-1473 20 mg; Test type: Superiority; p = 0.9542, Cochran-Mantel-Haenszel — P-value is shown for Cochran-Mantel Haenszel tests stratified by prior biologic failure and steroid use at baseline; Difference in Proportion = 0.00, 95% CI 2-sided [-0.104 to 0.110] — Difference in proportion estimates used Mantel-Haenszel stratum weights
Statistical Analysis 2: Comparison: Induction Period: Placebo vs Induction Period: TD-1473 80 mg; Test type: Superiority; p = 0.5863, Cochran-Mantel-Haenszel — P-value is shown for Cochran-Mantel Haenszel tests stratified by prior biologic failure and steroid use at baseline; Difference in Proportion = -0.03, 95% CI 2-sided [-0.126 to 0.071] — Difference in proportion estimates used Mantel-Haenszel stratum weights
Statistical Analysis 3: Comparison: Induction Period: Placebo vs Induction Period: TD-1473 200 mg; Test type: Superiority; p = 0.5408, Cochran-Mantel-Haenszel — P-value is shown for Conhran-Mantel Haenszel tests stratified by prior biologic failure and steroid use at baseline; Difference in Proportion = -0.03, 95% CI 2-sided [-0.131 to 0.069] — Difference in proportion estimates used Mantel-Haenszel stratum weights

4. Secondary Outcome: Phase 3 Maintenance: Number of Participants Who Demonstrated a Clinical Response by Adapted Mayo Score Components at mWeek 44
Description: Clinical response was defined as a reduction from baseline in adapted Mayo score of ≥ 2 points and ≥ 30% relative to baseline. It also required ≥ 1 reduction in the rectal bleeding subscore or an absolute subscore ≤ 1.
  The Adapted Mayo score was the sum of three components: rectal bleeding, stool frequency, and Mayo endoscopic subscore, each measured on a scale of 0-3 with higher scores reflecting higher severity.
  Participants with missing Week 44 values were imputed as non-responders.
Time Frame: Baseline to mWeek 44
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Period: Placebo | Maintenance Period: TD-1473 20 mg | Maintenance Period: TD-1473 80 mg | Maintenance Period: TD-1473 200 mg
Number analyzed (Participants) | 8 | 13 | 11 | 8
Participants | 5 | 5 | 8 | 6
Statistical Analysis 1: Comparison: Maintenance Period: Placebo vs Maintenance Period: TD-1473 20 mg; Test type: Superiority; p = 0.6656, Fisher Exact
Statistical Analysis 2: Comparison: Maintenance Period: Placebo vs Maintenance Period: TD-1473 80 mg; Test type: Superiority; p = 0.6424, Fisher Exact
Statistical Analysis 3: Comparison: Maintenance Period: Placebo vs Maintenance Period: TD-1473 200 mg; Test type: Superiority; p = 0.6199, Fisher Exact

5. Secondary Outcome: Phase 3 Maintenance: Number of Participants Who Demonstrated Endoscopic Remission by Adapted Mayo Score Components at mWeek 44
Description: Endoscopic remission was defined as an endoscopic subscore ≤ 1.
  Endoscopic subscore was measured using scale of 0-3, where higher numbers reflected greater severity.
Time Frame: mWeek 44
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Period: Placebo | Maintenance Period: TD-1473 20 mg | Maintenance Period: TD-1473 80 mg | Maintenance Period: TD-1473 200 mg
Number analyzed (Participants) | 9 | 13 | 11 | 8
Participants | 3 | 1 | 3 | 2
Statistical Analysis 1: Comparison: Maintenance Period: Placebo vs Maintenance Period: TD-1473 20 mg; Test type: Superiority; p = 0.2643, Fisher Exact
Statistical Analysis 2: Comparison: Maintenance Period: Placebo vs Maintenance Period: TD-1473 80 mg; Test type: Superiority; p = 1.0000, Fisher Exact
Statistical Analysis 3: Comparison: Maintenance Period: Placebo vs Maintenance Period: TD-1473 200 mg; Test type: Superiority; p = 1.0000, Fisher Exact

6. Secondary Outcome: Phase 3 Maintenance: Number of Participants Who Demonstrated Symptomatic Remission by Adapted Mayo Score Components at mWeek 44
Description: Symptomatic remission was defined as a stool frequency score ≤ 1 and a rectal bleeding subscore of 0.
  Stool frequency score and rectal bleeding score were each measured using scale of 0-3, where higher numbers reflected greater severity.
  Participants with missing Week 44 values were imputed as non-responders.
Time Frame: mWeek 44
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Period: Placebo | Maintenance Period: TD-1473 20 mg | Maintenance Period: TD-1473 80 mg | Maintenance Period: TD-1473 200 mg
Number analyzed (Participants) | 9 | 13 | 11 | 8
Participants | 5 | 7 | 7 | 5
Statistical Analysis 1: Comparison: Maintenance Period: Placebo vs Maintenance Period: TD-1473 20 mg; Test type: Superiority; p = 1.0000, Fisher Exact
Statistical Analysis 2: Comparison: Maintenance Period: Placebo vs Maintenance Period: TD-1473 80 mg; Test type: Superiority; p = 1.0000, Fisher Exact
Statistical Analysis 3: Comparison: Maintenance Period: Placebo vs Maintenance Period: TD-1473 200 mg; Test type: Superiority; p = 1.0000, Fisher Exact

ADVERSE EVENTS:
Time Frame: Induction Period: Up to Week 20 Maintenance Period: Up to Week 48
Description: The Safety analysis set included all participants who received at least one dose of study drug (TD-1473 or placebo).
Groups:
- Induction Period: Placebo: Participants who were randomized to receive once-daily administrations of placebo for 8 weeks during the Induction Period.
- Induction Period: TD-1473 20 mg: Participants who were randomized to receive once-daily administrations of 20 mg TD-1473 for 8 weeks during the Induction Period.
  Participants who did not achieve clinical response at Week 8 continued to receive 20 mg TD-1473 for 8 weeks in the Extended Induction Period.
- Induction Period: TD-1473 80 mg: Participants who were randomized to receive once-daily administrations of 80 mg TD-1473 for 8 weeks during the Induction Period.
  Participants who did not achieve clinical response at Week 8 continued to receive 80 mg TD-1473 for 8 weeks in the Extended Induction Period.
- Induction Period: Placebo to TD-1473 80 mg: Participants who were randomized to receive once-daily administrations of placebo for 8 weeks during the Induction Period.
  Participants who did not achieve clinical response at Week 8 received 80 mg TD-1473 for 8 weeks in the Extended Induction Period.
- Induction Period: TD-1473 200 mg: Participants who were randomized to receive once-daily administrations of 200 mg TD-1473 for 8 weeks during the Induction Period.
  Participants who did not achieve clinical response at Week 8 continued to receive 200 mg TD-1473 for 8 weeks in the Extended Induction Period.
- Maintenance Period: TD-1473 20 mg: Participants who achieved clinical response to a total of 8 weeks of TD-1473 induction therapy, either at Week 8 or Week 16, and were re-randomized to 20 mg TD-1473 for 44 weeks in the Maintenance Period.
- Maintenance Period: TD-1473 80 mg: Participants who achieved clinical response to a total of 8 weeks of TD-1473 induction therapy, either at Week 8 or Week 16, and were re-randomized to 80 mg TD-1473 for 44 weeks in the Maintenance Period.
- Maintenance Period: TD-1473 200 mg: Participants who achieved clinical response to a total of 8 weeks of TD-1473 induction therapy, either at Week 8 or Week 16, and were re-randomized to 200 mg TD-1473 for 44 weeks in the Maintenance Period.
Arm/Group | Induction Period: Placebo | Induction Period: TD-1473 20 mg | Induction Period: TD-1473 80 mg | Induction Period: Placebo to TD-1473 80 mg | Induction Period: TD-1473 200 mg | Maintenance Period: Placebo | Maintenance Period: TD-1473 20 mg | Maintenance Period: TD-1473 80 mg | Maintenance Period: TD-1473 200 mg
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/61 | 0/59 | 0/42 | 0/58 | 0/29 | 0/31 | 0/25 | 0/22
Serious Adverse Events (participants affected / at risk) | 4/61 | 4/61 | 2/59 | 3/42 | 4/58 | 1/29 | 2/31 | 2/25 | 1/22
Other Adverse Events (participants affected / at risk) | 7/61 | 11/61 | 9/59 | 4/42 | 14/58 | 6/29 | 14/31 | 5/25 | 1/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Induction Period: Placebo (N=61) | Induction Period: TD-1473 20 mg (N=61) | Induction Period: TD-1473 80 mg (N=59) | Induction Period: Placebo to TD-1473 80 mg (N=42) | Induction Period: TD-1473 200 mg (N=58) | Maintenance Period: Placebo (N=29) | Maintenance Period: TD-1473 20 mg (N=31) | Maintenance Period: TD-1473 80 mg (N=25) | Maintenance Period: TD-1473 200 mg (N=22)
Colitis ulcerative (Gastrointestinal disorders) | 2 | 3 | 1 | 1 | 2 | 0 | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cytomegalovirus colitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Liver abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestine operation (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Induction Period: Placebo (N=61) | Induction Period: TD-1473 20 mg (N=61) | Induction Period: TD-1473 80 mg (N=59) | Induction Period: Placebo to TD-1473 80 mg (N=42) | Induction Period: TD-1473 200 mg (N=58) | Maintenance Period: Placebo (N=29) | Maintenance Period: TD-1473 20 mg (N=31) | Maintenance Period: TD-1473 80 mg (N=25) | Maintenance Period: TD-1473 200 mg (N=22)
Colitis ulcerative (Gastrointestinal disorders) | 1 | 3 | 5 | 1 | 7 | 4 | 6 | 3 | 0
Nasopharyngitis (Infections and infestations) | 1 | 6 | 0 | 0 | 4 | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 2 | 1 | 2 | 1 | 3 | 0 | 1
Headache (Nervous system disorders) | 2 | 0 | 2 | 1 | 2 | 1 | 2 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 2 | 0 | 2 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was terminated early due to a company decision based on interim analysis results in TD-1473-0157. Therefore, the Phase 3 dose-confirming Induction Study was not conducted and the Maintenance Study was prematurely terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-05-14): https://cdn.clinicaltrials.gov/large-docs/43/NCT03758443/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-20): https://cdn.clinicaltrials.gov/large-docs/43/NCT03758443/SAP_001.pdf